CLINICAL TRIAL: NCT02643511
Title: Focal Low Dose Rate ( LDR) Brachytherapy: Hemi-ablative Treatment With LDR for Patients With Low and Low-tier Intermediate Risk Prostate Cancer
Brief Title: Hemiablative Focal Brachytherapy Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George Hospital, Australia (Other)
Responsible Party: Principal Investigator, Ana Fernandezots, Ana Fernandez Ots MD, St George Hospital, Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STGAF
Record Dates: First submitted 2015-07-22; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate biopsy,Hemiablative focal Brachytherapy (Experimental): This is a non-randomized, Phase II study examining the efficacy in terms of postimplant dosimetry (primary endpoint) as well as the secondary endpoints of QOL changes, toxicity, local control with post-treatment biopsy outcomes and comparison with historical whole-gland cohorts in men with early stage low volume prostate cancer treated with hemiablative focal brachytherapy
  Interventions: Radiation: Transperineal template guided mapping biopsy, multiparametric MRI, Hemiablative Focal Brachytherapy

INTERVENTIONS:
Radiation: Transperineal template guided mapping biopsy, multiparametric MRI, Hemiablative Focal Brachytherapy — A re-staging transperineal template guided mapping prostate biopsy as currently performed at participating institutions. Hemiablative Focal brachytherapy will be performed . The affected half of the prostate will be targeted with the prescription dose and receive 145 Gy of Iodine-125 (I-125). A postimplant dosimetry will be performed 30 days after procedure. The quality-of-life assessment will focus on erectile function, urinary function, bowel function, and general health related quality of life. The patients will complete this assessment at baseline and then 4 weeks, 6 months, 12 months, 20 months, 24 months, 32 months and 36 months after treatment. A second transperineal biopsy will be performed 36 months after the implant.

SUMMARY:
Whole gland LDR brachytherapy has been a well established modality of treating low risk prostate cancer. Treatment in a focal manner has the advantages of reduced toxicity to surrounding organs.

AIM: To determine the utility of focal LDR brachytherapy in form of hemiablative treatment for localized prostate cancer demonstrating the feasibility of the delivery of the prescription dose to the half of the prostate in terms of meeting standard dosimetric parameters while respecting same or lower tolerance doses of adjacent normal organs.

To determine acute and late rectal, urinary and sexual toxicity after this procedure.

To assess the change from baseline in QOL indicators at specific time intervals using validated international questionnaires [International Prostate Symptom Score ( IPSS), International Index of Erectile Function ( IIEF ), Expanded Prostate Cancer Index (EPIC)] after this treatment.

To evaluate the local tumour control in terms of biopsy outcomes after focal brachytherapy 36 months after the treatment.

To compare target coverage and relative doses to the rectum and the urethra for the same patient performing a hemigland treatment planning vs Whole gland treatment planning.

STUDY DESIGN: Multi-institution prospective trial to determine whether hemiablative treatment with LDR for prostate cancer is dosimetrically safe and feasible.This study will record data for 20 patients with ipsilateral with low and low tier intermediate risk disease.The study will record quality of life parameters in particular in terms of urinary, rectal and sexual function side effects.

INTERVENTION:

* Baseline Transperineal Template guided mapping prostate biopsy with >20 cores (not required if already performed)
* Multiparametric MRI within the 3 months prior to registration and at 18 & 36 months.
* Hemigland prostate region will be targeted with the prescription dose and receive 144 Gy of Iodine125 (I125).
* The quality of life assessment will focus on erectile function, urinary function, bowel function, and general health related quality of life
* Postimplant CT Planning day 30 after the implant for quality assurance.

MEASUREMENT OF ENDPOINTS :

Dosimetric parameters record, Toxicity and QOL evaluation forms, PSA follow up and biopsies at 36 months to assess local control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have histologically proven adenocarcinoma of the prostate.

  2. Patients must have low or low-tier intermediate prostate cancer
  * Low risk prostate cancer patients must have:

    * Clinical stage ≤ T2a,
    * Gleason score =6 and iPSA ≤ 10 ng/ml
    * < 25% cores positive, < 50 % cancer in each core involved
  * Low tier Intermediate risk patients may have:

    * Clinical stageT2a
    * Gleason score ≤ 3+4=7
    * PSA ≤ 10 ng/ml
    * < 25% cores positive, < 50 % cancer in each core

      3. Patients must be fit for general anesthetic. 4. Patients must have unilateral disease on biopsy 5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.

      6. Men ≥ 65 years of age with a life expectancy estimated to be >10 years. 7. Patients must have no contraindications to interstitial prostate brachytherapy.

      8. Patients on anticoagulant therapy must be able to stop therapy safely for at least 7 days.

      9. Patients must not have any contraindications to MRI 10. IPSS <=16

Exclusion Criteria:

1. Does not meet staging criteria for low risk or low tier intermediate risk prostate cancer
2. Bilateral prostatic disease
3. Prior hormonal therapy
4. Prior Transurethral resection or middle lobe resection
5. Recent IPSS>
6. Unfit for general anesthetic
7. MRI contraindicated
8. Unable to cease anticoagulant therapy
9. Life expectancy < 10 years
10. IPSS>16

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Optimal dosimetric parameters to target and organs at risk in day 30 postimplant dosimetry | 1month to 3 years
  Acceptable dosimetric parameters in Day 30 postimplant dosimetry as per brachytherapy guidelines

SECONDARY OUTCOMES:
Rates of acute and late toxicity assessed by CTCAE v4.0 | 6months to 10years
  Treatment related toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Change from baseline in QOL in Genitourinary aspect | 6 months to 10 years
  This will be assessed using the IPSS questionnaire
Change from baseline in QOL in the sexual aspect | 6 months to 10 years
  This will be assessed using the IIEF questionnaire
Change from baseline in QOL in the gastrointestinal aspect | 6 months to 10 years
  This will be assessed using the EPIC questionnaire
Local control as Negative prostate biopsy 36 months after the treatment | 3 years after treatment
Dosimetric parameters comparison between hemigland treatment vs Whole gland historical cohort | 6 months to 10 years
Grade of genitourinary and gastrointestinal toxicity assessed by CTCAE v4.0 comparison between hemigland treatment vs Whole gland historical cohort | 6 months to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- St George Hospital Cancer Care Centre, Kogarah, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Fernandez Ots A, Bucci J, Chin YS, Malouf D, Howie A, Enari KE. Hemiablative Focal Low Dose Rate Brachytherapy: A Phase II Trial Protocol. JMIR Res Protoc. 2016 Jun 13;5(2):e98. doi: 10.2196/resprot.5433. PMID 27296781